CLINICAL TRIAL: NCT05766579
Title: ElaStic-compressive Stockings at 21 mmHg and 32 mmHg Following Thermal Ablation of the Great Saphenous Vein.
Brief Title: Comparison Trial Between Elastic-compressive Stockings at 21 Versus 32 mmHg
Acronym: CALESSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Daniela Mazzaccaro, Medical Doctor and Researcher, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 41/int/2019
Record Dates: First submitted 2023-02-17; First posted 2023-03-13 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Vascular Surgical Procedures
Keywords: Stockings, Compression; Thermoablation; Radiofrequency; Saphenous Vein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- K1, 18-21 mmHg (Experimental): Use of elastic stockings at 18-21 mmHg after endovenous thermal ablation
  Interventions: Device: Elastic-compressive stockings
- K2, 23-32 mmHg (Experimental): Use of elastic stockings at 23-32 mmHg after endovenous thermal ablation
  Interventions: Device: Elastic-compressive stockings

INTERVENTIONS:
Device: Elastic-compressive stockings — Use of Elastic-compressive stockings at 21 mmHg and 32 mmHg.

SUMMARY:
Endovascular thermal ablation is currently considered as the best procedure for treating varicose veins thanks to its mini-invasiveness and the lowest rate of incidence of complications. At the end of the endovascular ablation procedure, the European Society of Vascular Surgery (ESVS) guidelines recommend the use of the compression stockings to reduce postoperative pain and the incidence of edema and thrombotic complications.

Despite this, the duration, type and degree of compression to be used, particularly after radiofrequency ablation procedures, remain a matter of debate. Furthermore, although the benefits of postoperative elastic compression therapy are well known, there is various evidence demonstrating how patients often experience poor comfort in wearing stockings, especially those with a higher degree of compression, which causes poor compliance with therapy. In light of all this, each center recommends the use of elastic compression stockings in the postoperative period with a degree of compression that varies, however, according to internal protocols.

There is currently no work in the literature that compares the advantages and disadvantages of using elastic compression stockings with a K2 versus K1 compression degree after radiofrequency ablative surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>18 years) suffering from varicose vein pathology of the lower limbs C2-3 class (varicose veins, edema) according to Clinic, Etiology, Anatomy, Pathophysiology (CEAP) classification, supported by incontinence of the great saphenous vein documented by Echo-Duplex study and candidates for thermal ablation by radiofrequency of the great vein saphenous vein with associated phlebectomy of the ipsilateral thigh and/or leg varices.

Exclusion Criteria:

* Patients who are minors (< 18 years old) or adults who have not given their consent to participate in the study.
* Presence of severe obliterating arterial disease of the lower limbs (ABI <0.5)
* Obesity (BMI >30)
* Varicose pathology of the lower limbs in C4-C6 class according to Clinic, Etiology, Anatomy, Pathophysiology (CEAP) classification (presence of:

lipodermatosclerosis/eczema and/or ulcers in progress and/or previous ulcers in the affected lower limb).

* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 3 days after surgery
  Evaluation of postoperative pain using the Visual Analogic pain Scale (1-10, being higher the pain the higher the value of the scale)
Postoperative Pain | 7 days after surgery
  Evaluation of postoperative pain using the Visual Analogic pain Scale (1-10, being higher the pain the higher the value of the scale)

SECONDARY OUTCOMES:
Lower limb edema | 3 days from intervention
  Evaluation of the circumference of the lower limb undergoing surgery in 3 points: 10 cm above the patella, at the level of the tibial tuberosity and 5 cm below the latter
Lower limb edema | 7 days from intervention
  Evaluation of the circumference of the lower limb undergoing surgery in 3 points: 10 cm above the patella, at the level of the tibial tuberosity and 5 cm below the latter
Lower limb edema | 30 days from intervention
  Evaluation of the circumference of the lower limb undergoing surgery in 3 points: 10 cm above the patella, at the level of the tibial tuberosity and 5 cm below the latter
Analgesic Drugs Use | 3 days from intervention
  Evaluation of the possible use of analgesic drugs for postoperative pain.
Analgesic Drugs Use | 7 days from intervention
  Evaluation of the possible use of analgesic drugs for postoperative pain.
Analgesic Drugs Use | 30 days from intervention
  Evaluation of the possible use of analgesic drugs for postoperative pain.
Discomfort | 3 days from intervention
  Evaluation of the discomfort caused to the patient by the use of stockings using the Aberdeen Varicose Veins Questionnaire .
Discomfort | 7 days from intervention
  Evaluation of the discomfort caused to the patient by the use of stockings using the Aberdeen Varicose Veins Questionnaire .
Discomfort | 30 days from intervention
  Evaluation of the discomfort caused to the patient by the use of stockings using the Aberdeen Varicose Veins Questionnaire .
Postoperative Complications | 3 days from intervention
  Evaluation of the incidence of postoperative complications
Postoperative Complications | 7 days from intervention
  Evaluation of the incidence of postoperative complications
Postoperative Complications | 30 days from intervention
  Evaluation of the incidence of postoperative complications
Evaluation of Quality of Life | 3 days from intervention
  Evaluation of the quality of life using a questionnaire
Evaluation of Quality of Life | 7 from intervention
  Evaluation of the quality of life using a questionnaire
Evaluation of Quality of Life | 30 days from intervention
  Evaluation of the quality of life using a questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S. Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
The authors of the study are the owners of all data collected and will commit to the publication of the data themselves unconditionally and in full.

REFERENCES:
- [Background] Wittens C, Davies AH, Baekgaard N, Broholm R, Cavezzi A, Chastanet S, de Wolf M, Eggen C, Giannoukas A, Gohel M, Kakkos S, Lawson J, Noppeney T, Onida S, Pittaluga P, Thomis S, Toonder I, Vuylsteke M, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Koncar I, Lindholt J, de Ceniga MV, Vermassen F, Verzini F, Document Reviewers, De Maeseneer MG, Blomgren L, Hartung O, Kalodiki E, Korten E, Lugli M, Naylor R, Nicolini P, Rosales A. Editor's Choice - Management of Chronic Venous Disease: Clinical Practice Guidelines of the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2015 Jun;49(6):678-737. doi: 10.1016/j.ejvs.2015.02.007. Epub 2015 Apr 25. No abstract available. PMID 25920631
- [Background] Onida S, Lane TR, Davies AH. Phlebectomies: to delay or not to delay? Phlebology. 2012 Apr;27(3):103-4. doi: 10.1258/phleb.2012.011130. No abstract available. PMID 22457169
- [Background] Huang TW, Chen SL, Bai CH, Wu CH, Tam KW. The optimal duration of compression therapy following varicose vein surgery: a meta-analysis of randomized controlled trials. Eur J Vasc Endovasc Surg. 2013 Apr;45(4):397-402. doi: 10.1016/j.ejvs.2013.01.030. Epub 2013 Feb 19. PMID 23433496
- [Background] Reich-Schupke S, Feldhaus F, Altmeyer P, Mumme A, Stucker M. Efficacy and comfort of medical compression stockings with low and moderate pressure six weeks after vein surgery. Phlebology. 2014 Jul;29(6):358-66. doi: 10.1177/0268355513484142. Epub 2013 May 3. PMID 23563646
- [Background] Ye K, Wang R, Qin J, Yang X, Yin M, Liu X, Jiang M, Lu X. Post-operative Benefit of Compression Therapy after Endovenous Laser Ablation for Uncomplicated Varicose Veins: A Randomised Clinical Trial. Eur J Vasc Endovasc Surg. 2016 Dec;52(6):847-853. doi: 10.1016/j.ejvs.2016.09.005. Epub 2016 Oct 17. PMID 27760697
- [Background] Bakker NA, Schieven LW, Bruins RM, van den Berg M, Hissink RJ. Compression stockings after endovenous laser ablation of the great saphenous vein: a prospective randomized controlled trial. Eur J Vasc Endovasc Surg. 2013 Nov;46(5):588-92. doi: 10.1016/j.ejvs.2013.08.001. Epub 2013 Sep 5. PMID 24012465
- [Background] Cavezzi A, Mosti G, Colucci R, Quinzi V, Bastiani L, Urso SU. Compression with 23 mmHg or 35 mmHg stockings after saphenous catheter foam sclerotherapy and phlebectomy of varicose veins: A randomized controlled study. Phlebology. 2019 Mar;34(2):98-106. doi: 10.1177/0268355518776127. Epub 2018 May 12. PMID 29754530
- [Background] El-Sheikha J, Carradice D, Nandhra S, Leung C, Smith GE, Wallace T, Campbell B, Chetter IC. A systematic review of the compression regimes used in randomised clinical trials following endovenous ablation. Phlebology. 2017 May;32(4):256-271. doi: 10.1177/0268355516648497. Epub 2016 May 12. PMID 27178404
- [Background] Weiss RA, Duffy D. Clinical benefits of lightweight compression: reduction of venous-related symptoms by ready-to-wear lightweight gradient compression hosiery. Dermatol Surg. 1999 Sep;25(9):701-4. doi: 10.1046/j.1524-4725.1999.99064.x. PMID 10491060
- [Background] Benigni JP, Sadoun S, Allaert FA, Vin F. Efficacy of Class 1 elastic compression stockings in the early stages of chronic venous disease. A comparative study. Int Angiol. 2003 Dec;22(4):383-92. PMID 15153823
- [Background] Liu R, Lao TT, Kwok YL, Li Y, Ying MT. Effects of graduated compression stockings with different pressure profiles on lower-limb venous structures and haemodynamics. Adv Ther. 2008 May;25(5):465-78. doi: 10.1007/s12325-008-0058-2. PMID 18523736
- [Background] El-Sheikha J, Carradice D, Nandhra S, Leung C, Smith GE, Campbell B, Chetter IC. Systematic review of compression following treatment for varicose veins. Br J Surg. 2015 Jun;102(7):719-25. doi: 10.1002/bjs.9788. Epub 2015 Apr 2. PMID 25833417
- [Background] Garratt AM, Macdonald LM, Ruta DA, Russell IT, Buckingham JK, Krukowski ZH. Towards measurement of outcome for patients with varicose veins. Qual Health Care. 1993 Mar;2(1):5-10. doi: 10.1136/qshc.2.1.5. PMID 10132081
- [Background] Krasznai AG, Sigterman TA, Troquay S, Houtermans-Auckel JP, Snoeijs M, Rensma HG, Sikkink C, Bouwman LH. A randomised controlled trial comparing compression therapy after radiofrequency ablation for primary great saphenous vein incompetence. Phlebology. 2016 Mar;31(2):118-24. doi: 10.1177/0268355514568658. Epub 2015 Jan 23. PMID 25616874